CLINICAL TRIAL: NCT05643872
Title: A Multicenter Open-Label Treatment Study Evaluating the Safety and Pharmacokinetics of QTORIN Rapamycin 3.9% Anhydrous Gel in the Treatment of Adults With Pachyonychia Congenita
Brief Title: A Study Evaluating the Safety and Pharmacokinetics of QTORIN Rapamycin 3.9% Anhydrous Gel in the Treatment of Adults With Pachyonychia Congenita
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Palvella Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALV-08
Record Dates: First submitted 2022-11-08; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Pachyonychia Congenita
MeSH Terms: conditions — Pachyonychia Congenita

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PTX-022 (Experimental)
  Interventions: Drug: PTX-022

INTERVENTIONS:
Drug: PTX-022 — QTORIN rapamycin 3.9% anhydrous gel

SUMMARY:
PALV-08 is a multicenter, open-label treatment (OLT) study enrolling adults with Pachyonychia Congenita (PC) with genotyped keratin mutations KRT6A, KRT6B, KRT6C or KRT16 who were previously enrolled in the PALV-05 (VAPAUS) trial.

The purpose of this OLT study is to investigate the safety of long term exposure and pharmacokinetics (PK) of QTORIN rapamycin 3.9% anhydrous gel or "PTX-022".

ELIGIBILITY:
Key Inclusion Criteria:

* Completed the PALV-05 (VAPAUS) study
* Agree to contraceptive use

Key Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Concomitant use of sirolimus or any sirolimus-containing medications (systemic or topical)
* Any significant concurrent condition that could adversely affect participation and/or the assessment of the safety and efficacy in the study
* Prior or planned treatment, including surgery or other medically necessary intervention deemed by the investigator that could adversely affect participation and/or the assessment of the safety and efficacy in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events | 6 months

SECONDARY OUTCOMES:
Pharmacokinetic parameters | Prior to dose, 12 hours and 24 hours
  AUC area under the sirolimus blood concentration-time profile

CONTACTS AND LOCATIONS:
Locations (1):
- Minnesota Clinical Study Center, New Brighton, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No